CLINICAL TRIAL: NCT02303262
Title: A Phase II Study of Mocetinostat Administered With Gemcitabine for Patients With Metastatic Leiomyosarcoma With Progression or Relapse Following Prior Treatment With Gemcitabine-Containing Therapy
Brief Title: SARC018: A Study of Mocetinostat and Gemcitabine in Patients With Metastatic Leiomyosarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sarcoma Alliance for Research through Collaboration (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SARC018
Record Dates: First submitted 2014-11-21; First posted 2014-11-27 (Estimated); Results first posted 2019-01-29 (Actual); Last update posted 2019-01-29 (Actual); Status verified 2018-11

CONDITIONS: Metastatic Leiomyosarcoma
MeSH Terms: conditions — Leiomyosarcoma | interventions — mocetinostat; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Mocetinostat and gemcitabine (Experimental): For each 21-day cycle, gemcitabine is administered on days 5 and 12 and mocetinostat is administered 3 days a week.
  Interventions: Drug: Mocetinostat; Drug: Gemcitabine

INTERVENTIONS:
Drug: Mocetinostat — Mocetinostat is taken orally at 70 mg/dose, 3 days per week, during cycle 1. Dose is increased to 90 mg starting at cycle 2.
Drug: Gemcitabine — Gemcitabine is administered via intravenous infusion at 1,000 mg/m2 at a rate of approximately 10 mg/m2/minute, on days 5 and 12 of every cycle.

SUMMARY:
This is an open-label, multi-center, Phase II trial studying the combination of mocetinostat and gemcitabine in patients who have previously demonstrated disease progression either while, or within six months after, receiving chemotherapy with a gemcitabine-based regimen.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Histologically documented leiomyosarcoma
* Prior systemic therapy with a gemcitabine containing regimen
* ECOG Performance Status of ≤ 1
* Measurable metastatic disease with a target lesion that has increased in size by 20% in maximal dimension either during or within six months after treatment with chemotherapy using a gemcitabine containing regimen
* Adequate organ function within 14 days of study entry
* Patients or their legal representative must be able to read (or have read to them), understand, and sign a written informed consent (approved by the institutional review board) within 14 days prior to start of treatment.

Exclusion Criteria:

* Concurrent, clinically significant, active malignancies (excluding basal cell carcinoma or cervical intraepithelial neoplasia [CIN] in situ or melanoma in situ) (Stage II portion only)
* Patients with baseline QTcF ≥ 480 msec
* Patients with uncontrolled concurrent illness, active infection requiring i.v. antibiotics, or uncontrolled infections, or a fever > 38.5°C on the day of scheduled dosing
* Patients with serious illnesses, medical conditions, or other medical history, including a prior history of pericarditis/pericardial effusion, or abnormal laboratory results, which, in the investigator's opinion, would be likely to interfere with a patient's participation in the study, or with the interpretation of the results
* Patients who have received any investigational drug within 28 days prior to Day 1 of study entry (an investigational drug is one for which there is no approved indication), or who are receiving concurrent treatment with other experimental drugs or anti-cancer therapy
* Pregnant or lactating women. Women of child-bearing potential (WOCBP) must have a negative serum pregnancy test documented within 72 hours prior to starting study drug or a urine pregnancy test shall be done on Day 1 of Cycle 1
* Women of child bearing potential and their partners must use an acceptable method of contraception while enrolled on this study, and for a period of 3 months following study drug treatment. Patients unwilling or unable to follow this guideline will be excluded. Investigators should follow their Institutional standard regarding acceptable methods of contraception.
* Known hypersensitivity to HDAC inhibitors or to any of the components of mocetinostat
* Known hypersensitivity to gemcitabine
* Any condition that will put the patient at undue risk or discomfort as a result of adherence to study procedures. For example, consider requirement to take mocetinostat with water and recommendation to avoid agents that increase gastric pH
* Any condition (e.g., known or suspected poor compliance, psychological instability, geographical location, etc) that, in the judgment of the investigator, may affect the patient's ability to sign the informed consent and undergo study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-11-12 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edwin Choy, MD, PhD, Principal Investigator — MGH, Dana Farber/Harvard Cancer Center; Shreyas Patel, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (5):
- United States (5):
  - Massachusetts General Hospital/Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Ohio State University, Columbus, Ohio
  - University of Texas MD Anderson Cancer Center, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Mocetinostat and Gemcitabine
Started | 20
Completed | 18
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Mocetinostat and Gemcitabine
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 17
  >=65 years | 3
Age, Continuous [Mean (Full Range); unit: years] | 56.8 [39 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 15
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Response Rate (Per RECIST 1.1)
Description: Response rate (CR or PR) will be calculated by the number of patients achieving a response divided by the number of patients having been evaluated for response. Per Response Evaluation Criteria in Solid Tumors (RECIST): Complete Response (CR) is the disappearance of all target lesions; Partial Response (PR) is at least a 30% decrease in the sum of longest diameters of all target lesions.
Time Frame: 27 months
Measure: Count of Participants; unit: Participants
Arm/Group | Mocetinostat and Gemcitabine
Number analyzed (Participants) | 18
Participants | 1

2. Secondary Outcome: Duration of Response
Description: The duration of objective response will be measured from the time measurement criteria are first met until disease progression is objectively documented.
Time Frame: 27 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Mocetinostat and Gemcitabine
Number analyzed (Participants) | 18
months | 2 [1.5 to 3.1]

3. Secondary Outcome: Progression Free Survival (PFS)
Description: Progression free survival is defined as the time from treatment initiation to the earlier date of assessment of objective progression or death by any cause in the absence of progression. Progression Free Survival (PFS) is defined as the time from treatment initiation to the earlier date of assessment of objective progression or death by any cause in the absence of progression. Progression will be assessed by RECIST v. 1.1.
Time Frame: 27 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Mocetinostat and Gemcitabine
Number analyzed (Participants) | 18
months | 2.0 [1.5 to 3.1]

ADVERSE EVENTS:
Time Frame: through study completion, an average of 3 months
Arm/Group | Mocetinostat and Gemcitabine
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 12/20
Other Adverse Events (participants affected / at risk) | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mocetinostat and Gemcitabine (N=20)
Anemia (Blood and lymphatic system disorders) | 2 (2)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Failure to thrive (General disorders) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Fever (General disorders) | 2 (2)
Hypotension (Vascular disorders) | 1 (1)
Mucositis (General disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Neutropenia (Investigations) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Pain (General disorders) | 2 (2)
Pericardial effusion (Cardiac disorders) | 1 (1)
Platelet count decreased (Investigations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mocetinostat and Gemcitabine (N=20)
Absolute neutrophil count decreased (Investigations) | 1 (3)
Achy (General disorders) | 1 (1)
Acid reflux (Gastrointestinal disorders) | 2 (2)
Alanine Aminotransferase increased (Investigations) | 1 (2)
Alkaline phosphatase increased (Investigations) | 2 (3)
Anemia (Blood and lymphatic system disorders) | 8 (28)
Anorexia (Metabolism and nutrition disorders) | 6 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Bruising (Injury, poisoning and procedural complications) | 1 (1)
Burping (Gastrointestinal disorders) | 1 (1)
Calf tenderness/burning (Musculoskeletal and connective tissue disorders) | 1 (1)
Chills (General disorders) | 2 (2)
Cord compression (General disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Creatinine increased (Investigations) | 1 (2)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 4 (8)
Dizziness (Nervous system disorders) | 2 (3)
Dry mouth (Gastrointestinal disorders) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 4 (4)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Ejection fraction decreased (Investigations) | 1 (1)
Elevated LFTs (Investigations) | 1 (1)
Erythematous neck rash (Skin and subcutaneous tissue disorders) | 1 (1)
Facial acne (Skin and subcutaneous tissue disorders) | 1 (1)
Fatigue (General disorders) | 12 (22)
Fever (General disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
GGT increased (Investigations) | 1 (1)
Headache (Nervous system disorders) | 2 (2)
Hypertension (Vascular disorders) | 2 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (2)
Insomnia (Psychiatric disorders) | 4 (4)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sciatic pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Lymphocyte count decreased (Investigations) | 2 (5)
Malaise (General disorders) | 1 (1)
Memory impairment (Nervous system disorders) | 1 (1)
Muscle cramps (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Nasal irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 8 (12)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Neck stiffness (Musculoskeletal and connective tissue disorders) | 1 (1)
Neutrophil count decreased (Investigations) | 8 (18)
Night sweats (General disorders) | 1 (1)
Sore nostril (Skin and subcutaneous tissue disorders) | 1 (1)
Pain (General disorders) | 2 (3)
Thigh pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Paresthesia (Nervous system disorders) | 1 (1)
Pericardial tamponade (Cardiac disorders) | 1 (1)
Pericarditis (Cardiac disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (3)
Pharyngitis (Infections and infestations) | 1 (1)
Platelet count decreased (Investigations) | 6 (16)
Powerport soreness (Injury, poisoning and procedural complications) | 1 (1)
Pruritic rash (Skin and subcutaneous tissue disorders) | 1 (1)
Pulmonary embolism (Blood and lymphatic system disorders) | 1 (1)
QTCF elevated (Cardiac disorders) | 1 (1)
Fungal infection (Infections and infestations) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 1 (1)
Right sided chest pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Sharp left sided pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Shoulder pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (1)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Thrush (Infections and infestations) | 1 (1)
Ventricular arrhythmia (Cardiac disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 5 (8)
Weight loss (Investigations) | 1 (1)
White blood cell decreased (Investigations) | 4 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No